CLINICAL TRIAL: NCT05958368
Title: The Effects of Hass Avocados on Glycemic Control in Persons With Type 2 Diabetes: A Randomized Controlled Crossover Trial
Brief Title: Assessing the Value of Avocados on Glycemic Control in Type 2 Diabetes
Acronym: AVOCADO-T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Prachi Singh (Unknown); Frank L. Greenway (Unknown); Robbie A. Beyl (Unknown)
Responsible Party: Principal Investigator, John Apolzan, Associate Professor-Research, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2023-033
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Insulin; Fructosamine; C-Reactive Protein; Glucose; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This study utilizes a randomized crossover design with each period/treatment being approximately 5 weeks. Participants will be randomized to either Hass Avocado or other fruit(s) consumption groups. The treatments will be isocaloric as will the Hass Avocado vs. the other fruit(s). All subjects will consume a diet provided by the metabolic research kitchen. The diet will be matched on energy (kcal).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and outcome assessors will be blinded to study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avocado (Experimental): Participants will consume 1 Hass avocado a day.
  Interventions: Other: Avocado
- Other Fruit(s) (Active Comparator): Participants in the other fruit arm will receive other fruits.
  Interventions: Other: Other Fruit(s)

INTERVENTIONS:
Other: Avocado — The Hass Avocado group will consume 7 avocados a week (1 / day; ~240 kcals/d).
  Other Names: Hass Avocado
  Arms: Avocado
Other: Other Fruit(s) — The other fruits group will consume fruit(s) matched to the avocado in energy and form (i.e., solid fruit).
  Other Names: Raisins, Cantaloupe(s), Figs, Pineapple(s), Grapes, Bananas
  Arms: Other Fruit(s)

SUMMARY:
The objective of this study is to assess the effects of Hass Avocados on glycemic control. The investigators hypothesize that Hass Avocado consumption will reduce fasting blood sugar compared to an isocaloric amount of other fruit during controlled feeding.

ELIGIBILITY:
Inclusion Criteria:

* Participant reported diagnosis of Type 2 diabetes
* HbA1c between 5.7%-11% (inclusive) and / or fasting blood glucose of ≥ 100 mg/dL
* BMI 27-50 kg/m2 (inclusive)
* Age range - 18 - 65 years (inclusive)
* On stable regimen of all medications (including diabetes) for at least 3 months (brief regimens of medications such as antibiotics, steroids, etc. are permitted)
* Willing to follow all requirements of study protocol including blood draws
* Under the care of a physician who will be responsible for managing the subject's diabetes
* Willing to give release to provide their treating MD with information about the trial

Exclusion Criteria:

* Not willing or unable to consume study foods including avocados
* Participation in a weight control program within the past 3 months or weight loss of ≥ 5 kg in the previous 3 months
* Taking prescription or OTC weight loss medications within last 4 weeks
* History of a surgical procedure for weight loss in last 5 years (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve)
* History of major surgery within three months of enrollment
* Type 1 diabetes, insulin dependent type 2 diabetes, thiazolidinediones (including rosiglitazone and pioglitazone)
* Renal insufficiency consisting of potassium over 5.5 (mmol/L) on a non-hemolyzed specimen, or a creatinine over 2.5 mg/dL
* Bilirubin over 3 (mg/dL) or an albumin less than 3 (g/dL)
* ALT > 3 (IU/L) times the upper limit of normal (normal range is 7-56)
* Evidence of more than 1 severe hypoglycemic event (episode requiring emergency medical services) in the past 12 months, unless the participant's treating physician provides written clearance for participation.
* Those on higher doses of diuretics (furosemide 40mg or higher or comparable)
* Unstable heart disease (an ongoing workup or treatment for a cardiac symptom such as unstable angina, coronary ischemia)
* Presence of implanted cardiac defibrillator
* Blood pressure ≥180/100 mm Hg. If a potential participant has a BP above the inclusion criteria it is acceptable to re-test this potential participant within one week of the original test.
* Thyroid disease for which the participant is untreated or has had treatment changed within the last 6 months. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable
* Uncontrolled gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea, or active gallbladder disease
* Current cancer or cancer treatment, or a history of cancer or cancer treatment within the last 3 years. Persons with successfully resected non-melanoma carcinoma of the skin may be enrolled.
* Dementia, psychiatric illness, or substance abuse that may interfere with adherence (e.g., illness that is currently unstable or resistant to first-line therapy; substance abuse in the past year)
* Women who are pregnant, lactating, trying to become pregnant or unwilling to use an effective means of birth control
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and unwilling to stop intake during study participation
* Participation in another clinical trial within 30 days prior to enrollment
* Any other condition or factor which in the opinion of the study physician or investigator makes it inadvisable for the candidate to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose | Week 5 - Week 0
  the primary outcomes are based on within subject concentration change scores

SECONDARY OUTCOMES:
Fasting Insulin | Week 5 - Week 0
  within subject concentration change scores
Fructosamine | Week 5 - Week 0
  within subject concentration change scores
Glycated Albumin | Week 5 - Week 0
  within subject concentration change scores

OTHER OUTCOMES:
Blood Glucose | Week 5 - Week 0
  Continuous Glucose Monitoring
Glucose | Week 5 - Week 0
  Oral Glucose Tolerance Test (OGTT)
Insulin | Week 5 - Week 0
  Oral Glucose Tolerance Test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be requested. The PI and sponsor will be notified. The proposed research question must be included. All IPD that underlie results in a publication after a DTA with the institution.